CLINICAL TRIAL: NCT04670354
Title: Differential Diagnosis and Cause-specific Treatment During OHCA - a Prospective Feasibility Study
Brief Title: Differential Diagnosis and Cause-specific Treatment During OHCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jouni Nurmi, MD, docent, specialist in anesthesiology and intensive care, Helsinki University Central Hospital
Other Study IDs: HUS-247-2020-9
Record Dates: First submitted 2020-11-16; First posted 2020-12-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: out of hospital cardiac arrest; differential diagnosis; prospective; ultrasound; blood gas analyse
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Differential diagnosis: ultrasound, blood gas analyse combined with examination of the patient and environment is used during Out Of Hospital Cardiac Arrest (OHCA) to screen possible underlying cause of cardiac arrest. Helicopter Emergency Medical Service (HEMS) in Helsinki has unraveled a protocol for performing differential diagnosis during OHCA. Our study aim is to test the feasibility of this protocol. Our study is a prospective medical record based study. The anesthesiologist operating in the HEMS unit fills a form after encounter of OHCA. Questioners focus on how long did execution of the protocol take, and the cause if the protocol was not completed.

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic out-of-hospital cardiac arrest encountered by the helicopter emergency medical services team

Exclusion Criteria:

* return of spontaneous circulation before HEMS crew arrival
* termination of resuscitation attempt before HEMS crew arrival

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-traumatic out-of-hospital cardiac arrest patients encountered by the helicopter emergency medical services.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-06-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Successful execution of differential diagnosis protocol | 60 minutes
  Successful and all-inclusive execution of the following items during cardiopulmonary resuscitation: ultrasound examination, arterial blood gas analyze, clinical examination, obtaining structured history from next of kin and searching of the environment.

SECONDARY OUTCOMES:
Rate of cause-specific treatment during resuscitation | 60 minutes
  Any therapy given as a treatment of presumed reversible cause of a cardiac arrest (excluding chest-compressions, ventilation, airway management, oxygen, epinephrine, amiodarone and defibrillation)
Time needed to complete the differential diagnostics protocol | 60 minutes
  Delay from patient encountered by the prehospital critical care physician to the all diagnostics performed (during cardiopulmonary resuscitation)

CONTACTS AND LOCATIONS:
Locations (1):
- FinnHEMS 10, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided